CLINICAL TRIAL: NCT04447781
Title: A Phase I/IIa, Dose-Ranging Trial to Evaluate Safety, Tolerability and Immunogenicity of INO-4800, a Prophylactic Vaccine Against SARS-CoV-2, Administered Intradermally Followed by Electroporation in Healthy Volunteers
Brief Title: Safety, Tolerability and Immunogenicity of INO-4800 Followed by Electroporation in Healthy Volunteers for COVID19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other); Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: IVI COVID19-001
Record Dates: First submitted 2020-06-16; First posted 2020-06-25 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Coronavirus Infection; SARS-CoV 2
Keywords: Coronavirus Infection; SARS-CoV 2; INO-4800
MeSH Terms: conditions — Coronavirus Infections | interventions — reluscovtogene ralaplasmid; Buffers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part A: Open Label Part B: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Group 1 (Part A) (Experimental): * Number of Subjects: 20 subjects
  * ID Injection of INO-4800 1mg/dose + EP using CELLECTRA® 2000 (dosing at Day 0 and Week 4)
  Interventions: Biological: INO-4800; Device: CELLECTRA® 2000
- Group 2 (Part A) (Experimental): * Number of Subjects: 20 subjects
  * ID Injection of INO-4800 2mg/dose + EP using CELLECTRA® 2000 (dosing at Day 0 and Week 4)
  Interventions: Biological: INO-4800; Device: CELLECTRA® 2000
- Group 3 (Part B) (Experimental): * Number of Subjects: 90 subjects
  * ID Injection of INO-4800 1mg or 2mg/dose + EP using CELLECTRA® 2000 (dosing at Day 0 and Week 4)
  Interventions: Biological: INO-4800; Device: CELLECTRA® 2000
- Group 4 (Part B, Placebo) (Placebo Comparator): * Number of Subjects: 30 subjects
  * ID Injection of Placebo (SSC) 1mg or 2mg/dose + EP using CELLECTRA® 2000 (dosing at Day 0 and Week 4)
  Interventions: Device: CELLECTRA® 2000; Other: Saline-sodium citrate (SSC) buffer

INTERVENTIONS:
Biological: INO-4800 — - Manufacturer: Inovio Pharmaceuticals Inc.
  Arms: Group 1 (Part A); Group 2 (Part A); Group 3 (Part B)
Device: CELLECTRA® 2000 — - Manufacturer: Inovio Pharmaceuticals Inc.
Other: Saline-sodium citrate (SSC) buffer — - Manufacturer: Inovio Pharmaceuticals Inc.
  Other Names: Placebo
  Arms: Group 4 (Part B, Placebo)

SUMMARY:
This is a phase I/IIa trial to evaluate the safety, tolerability and immunological profile of INO-4800 administered by intradermal (ID) injection followed by electroporation (EP) using the CELLECTRA® 2000 device in healthy adults aged 19 to 64 years in Republic of Korea. INO- 4800 contains the plasmid pGX9501, which encodes for the full length of the Spike glycoprotein of SARS-CoV-2. The primary objective of this trial is to evaluate the tolerability, safety, and immunogenicity of INO-4800 administered by ID injection followed by EP in healthy adults in the Part A and Part B. Enrollment into Part A, and Part B will proceed sequentially.

DETAILED DESCRIPTION:
[Part A] Part A is open-label, dose-ranging study, enrolling total of 40 subjects. Part A is divided into two arm, low dose (Group 1) and high dose (Group 2). The subjects will be contacted by telephone to report adverse events or other reactions the day following the first vaccination. Once these first five subjects in Group 1 complete the Week 1 visit, all available clinical laboratory and adverse event data will be reviewed by the Data Safety Monitoring Board (DSMB). Further enrollment into Group 1 will be paused during this DSMB review. If DSMB determines there are no safety findings judged to be of clinical concern and no dose limiting toxicities nor any stopping events observed, enrollment will be opened for the remaining subjects in Group 1. Once Group 1 enrollment is completed [i.e., 20 total subjects enrolled], Group 2 will open to enrollment. Daily safety assessment of all enrolled subjects will be supported by the Study Medical Monitor on an ongoing basis while the first five subjects are being enrolled, if needed. The subjects will be contacted by telephone to report adverse events or other reactions the day following the first vaccination. Once the first five subjects Group 2 complete the Week 1 visit, all available clinical laboratory and adverse event data from these first five subjects, along with the safety data from subjects in Group 1, will be reviewed by the DSMB. However, enrollment may continue while this DSMB review is conducted, without any pause to enrollment of the remaining subjects in Group 2.

Once all subjects in Part A Group 1 and Group 2 complete the Week 8 visit, all available clinical laboratory, adverse event, immunogenicity data from all subjects will be reviewed by the DSMB. The DSMB will additionally review serious adverse events (SAEs) and adverse events of special interest (AESIs) date throughout the study. With DSMB's recommendation, the optimal dose for Part B will be selected by the Sponsor based on the following criteria which may be adjusted over the course of the study. Percentage immunogenic seroconversionRelative immunogenicity between INO-4800 Study Arms (Low dose vs. High dose)Safety profile of each INO-4800 Study Arms (Low dose vs. High dose). All subjects will be followed for 48 weeks following the 2nd vaccination. Week 52 will be the End of Study (EOS) visit.

[Part B] Part B is divided into two arm, IP Arm (Group 3) and Placebo Arm (Group 4). Part B will be randomized, double-blind, placebo-controlled trial, enrolling 60 subjects in IP arm, and 20 subjects in Placebo arm in 19-50 age group, and 30 subjects in IP arm, and 10 subjects in Placebo arm in 51-64 age group, for total of 90 subjects in IP arm, and 30 subjects in Placebo arm. At dosing visit, subjects will be randomized to either Group 3 or Group 4. The subjects will be contacted by telephone to report adverse events or other reactions the day following the first vaccination. DSMB review of safety findings will be performed according to the DSMB charter. All subjects will be followed for 48 weeks following the 2nd vaccination. Week 52 will be the End of Study (EOS) visit.Should the criteria for any dose limiting toxicity or stopping rule be met, at any time, further enrollment and administration of INO-4800 will be paused for further evaluation. The Sponsor will consult the DSMB, if needed, to determine whether to enroll and/or dose the remainder of the subjects. All subjects will be followed for 48 weeks following the 2nd vaccination. Week 52 will be the End of Study (EOS) visit.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate with investigator, and to provide informed consent and have signed Informed Consent Form (ICF) prior to screening procedures
* Adults aged 19 to 50 years (for Part A) or aged 19 to 64 (for Part B)
* Judged to be healthy by the Investigator on the basis of medical history, physical examination and vital signs performed at Screening
* Able and willing to comply with all study procedures
* Screening laboratory results within normal limits for testing laboratory or deemed not clinically significant by the Investigator
* Negative serological tests for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody and Human Immunodeficiency Virus (HIV) antibody or rapid test at screening
* Screening ECG and Chest X-ray deemed by the Investigator as having no clinically significant findings (e.g. Wolff-Parkinson-White syndrome);
* Must meet one of the following criteria with respect to reproductive capacity:

  a. Women who are post-menopausal as defined by spontaneous amenorrhea for ≥ 12 months b. Surgically sterile or have a partner who is sterile (i.e., vasectomy in males or tubal ligation, absence of ovaries and/or uterus in females). In the case of vasectomy, subjects should wait six (6) months post-vasectomy prior to enrolling c. Use of medically effective contraception with a failure rate of < 1% per year when used consistently and correctly from screening until 3 months following last dose. Acceptable methods include (but not limited to): c-1. hormonal contraception including implants, injections or oral c-2. two barrier methods, e.g., condom and cervical cap (with spermicide) or diaphragm (with spermicide)

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant or father children within the projected duration of the trial starting with the screening visit until 3 months following last dose
* Positive serum pregnancy test during screening or positive urine pregnancy test prior to dosing
* Is currently participating in or has participated in a study with an investigational product within 6 months preceding Day 0
* Receipt of an investigational product for prophylaxis or treatment of COVID-19, MERS or SARS
* Body mass index (BMI) <18 or >30
* Current or history of the following medical conditions:

  1. Respiratory diseases (e.g., asthma, chronic obstructive pulmonary disease);
  2. Hypertension, resting systolic blood pressure >150 mm Hg or a diastolic blood pressure >95 mm Hg
  3. Malignancy within 5 years of screening
  4. Cardiovascular diseases (e.g., myocardial infarction, congestive heart failure, cardiomyopathy or clinically significant arrhythmias)
  5. Diabetes mellitus
  6. Use of immunoglobulin or blood products in last 6 months
  7. History of severe allergic reaction or anaphylaxis after immunization
* Immunosuppression as a result of underlying illness or treatment including:

  1. Primary immunodeficiencies
  2. Long term use (≥7 days) of oral or parenteral glucocorticoids at a dose of ≥20 mg/day of prednisone equivalent (use of inhaled, topical, nasal, otic, and ophthalmic corticosteroids are allowed)
  3. Current or anticipated during clinical trial use of disease modifying doses of anti-rheumatic drugs (e.g., azathioprine, cyclophosphamide, cyclosporine, methotrexate) and biologic disease modifying drugs such as TNF-α inhibitors (e.g., infliximab, adalimumab or etanercept)
  4. History of solid organ or bone marrow transplantation
  5. Any prior history of other clinically significant immunosuppressive or clinically diagnosed autoimmune disease that may jeopardize the safety of the subject or require therapy that would interfere with study assessments or endpoint evaluation, or otherwise impact the validity of the study results.
* Fewer than two acceptable sites available for ID injection and EP considering the deltoid and anterolateral quadriceps muscles. The following are unacceptable sites:

  1. Tattoos, keloids or hypertrophic scars located within 2 cm of intended administration site
  2. Implantable-Cardioverter-defibrillator (ICD) or pacemaker (to prevent a life-threatening arrhythmia) that is located ipsilateral to the deltoid injection site (unless deemed acceptable by a cardiologist)
  3. Any metal implants or implantable medical device within the electroporation site
* Prisoners or subjects who are compulsorily detained (involuntary incarceration)
* Reported active drug or alcohol or substance abuse or dependence.
* Current smoker or vaper (use of cigarette or e-cigarette at least once in last 30 days)
* Healthcare worker who may provide medical care to SARS-CoV-2 cases or occupationally in high risk for SARS-CoV-2 exposure during the study period
* Other condition deemed ineligible for the study at the discretion of investigator
* Employee of the study center directly involved with the proposed study or with study investigators
* Previously been laboratory-confirmed as SARS-CoV-2 infection or determined to be a close-contact of SARS-CoV-2 confirmed case by public health authorities (for Part A only)

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measures | Baseline up to Week 52
  * Percentage of participants with seroconversion of SARS-CoV-2 Spike glycoprotein antigen-specific antibody titers from baseline by binding assays [Immunogenicity]
  * Incidence of adverse events among participants during the study period [Safety and Tolerability]
  * Percentage of Participants with Administration (Injection) Site Reactions [Safety and Tolerability]
  * Incidence of Adverse Events of Special Interest (AESIs) among participants during the study period [Safety and Tolerability]

CONTACTS AND LOCATIONS:
Overall Officials: Myoung-don Oh, MD, Principal Investigator — Seoul National University Hospital; Eu Suk Kim, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries and all collected IPD will be anonymized and may be made available upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Anonymous IPD may be shared following or during the publication of summary data. Archival data may be accessed for up to 3 years following the end of the study.
Access Criteria: Those who request the anonymous IPD must provide a plan of study explaining how the data will be used. Requests may be sent to the Central Contact Person. Requests will be reviewed based on the potential for the planned use of the IPD for advancing scientific knowledge and theory.